CLINICAL TRIAL: NCT01830842
Title: Acute and Chronic Nicotine Modulation of Reinforcement Learning
Acronym: NicLearning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00043890
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Nicotine Addiction
Keywords: Nicotine; Smoking; Cigarettes; Reinforcement Learning; fMRI
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Tobacco Use Cessation Devices; Natural Family Planning Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine, placebo (Placebo Comparator): Nonsmokers will be measured following a nicotine polacrilex lozenge (2mg) on one occasion and placebo on another occasion.
  Interventions: Drug: Nicotine polacrilex; Drug: Placebo
- Nicotine withdrawal or satiety (Other): Smokers will be measured in a normal satiated condition and following 24-hours of smoking abstinence
  Interventions: Other: satiety; Other: abstinence

INTERVENTIONS:
Drug: Nicotine polacrilex — nonsmokers will be measured following nicotine administration
  Other Names: nicotine condition
  Arms: Nicotine, placebo
Drug: Placebo — nonsmokers will be measured following placebo administration
  Other Names: placebo condition
  Arms: Nicotine, placebo
Other: satiety — smokers will be measured in a smoking satiated condition
  Other Names: smoking satiated condition
  Arms: Nicotine withdrawal or satiety
Other: abstinence — smokers will be measured following 24-hours of smoking abstinence
  Other Names: smoking abstinence condition
  Arms: Nicotine withdrawal or satiety

SUMMARY:
The purpose of this study is to use functional magnetic resonance imaging (fMRI) to investigate the acute and chronic effects of nicotine on motivational behavior and prediction error-related neural activation. Nonsmokers (n = 24) and smokers (n = 24) will undergo fMRI scans on two separate occasions while performing a decision-making task that will elicit prediction error signals in the mesocorticolimbic pathway of the brain. Nonsmokers will be scanned once following an acute dose of nicotine and once following placebo administration. Smokers will be scanned once following smoking as usual and once following 24-hours of smoking abstinence, in order to measure the effects of nicotine withdrawal. The study team hypothesizes that acute nicotine will increase the prediction error signal in nonsmokers compared to placebo, and that nicotine withdrawal will decrease the prediction error signal in smokers compared to the normal satiated condition. Furthermore, nonsmokers (during the placebo condition) will have greater prediction error activation than smokers (during the satiated condition). The results of this study will inform whether the initiation and maintenance of smoking behavior could be facilitated by the effects of nicotine on reinforcement learning.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all subjects:

1. generally healthy
2. between the ages of 18-55
3. right-handed

Inclusion criteria for nonsmokers:

1. smoked < 50 cigarettes of a brand delivering ≥ 0.5 mg nicotine (FTC method)
2. have not smoked in ≥ 6 months
3. afternoon expired CO concentration ≤ 5 ppm and/or morning urinary NicAlert < 100 ng/ml

Inclusion criteria for smokers

1. smoke ≥ 10 cigarettes/day of a brand delivering ≥ 0.5 mg nicotine (FTC method)
2. smoked ≥ 2 years
3. afternoon expired CO concentrations ≥ 10 ppm and/or morning urinary NicAlert > 100 ng/ml

Exclusion Criteria:

1. inability to attend all required experimental sessions
2. significant health problems (e.g., current and uncontrolled liver, lung, or heart problems, current or past seizure disorder, serious head trauma)
3. lifetime diagnosis of Axis I psychiatric disorders (e.g., depression, anxiety disorder, schizophrenia)
4. meet DSM-V criteria for past or current substance dependence other than nicotine
5. use of psychoactive medications as indicated by self-report
6. use of smokeless tobacco, nicotine replacement therapy, or desire to change smoking behavior while in the study
7. positive urine drug screen for illicit drugs or positive breath alcohol concentration
8. presence of conditions that would make MRI unsafe
9. having vision that cannot be corrected to 20/40
10. among women, nursing or a positive pregnancy test
11. inability to achieve learning criteria in training session

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-02; Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merideth A Addicott, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotine, Placebo | Nicotine Withdrawal or Satiety
Started | 30 | 24
Completed | 25 | 22
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine, Placebo | Nicotine Withdrawal or Satiety | Total
Number analyzed (Participants) | 30 | 24 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 24 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (11) | 35 (10) | 34 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 13 | 10 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 24 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Oxygen Level Dependent (BOLD) Signal in Dorsomedial Prefrontal Cortex
Description: The acute and chronic effects of nicotine on the blood oxygen level dependent signal will be measured using functional magnetic resonance imaging. Reward-cue related BOLD signal on an outcome expectation task.
Time Frame: Nonsmokers: post nicotine and post placebo. Smokers: 24 hours smoking abstinence or smoking satiety
Population: Subjects who did not follow MRI task instructions, or those with > 3 mm of movement, were excluded from the analyses.
Measure: Mean (Standard Deviation); unit: percentage of BOLD signal
Groups:
- Nonsmokers: Nonsmokers will be measured following a nicotine polacrilex lozenge (2mg) on one occasion and placebo on another occasion.
  Nicotine polacrilex: nonsmokers will be measured following nicotine administration
  Placebo: nonsmokers will be measured following placebo administration
- Smokers: Smokers will be measured in a normal satiated condition and following 24-hours of smoking abstinence
  satiety: smokers will be measured in a smoking satiated condition
  abstinence: smokers will be measured following 24-hours of smoking abstinence
Arm/Group | Nonsmokers | Smokers
Number analyzed (Participants) | 23 | 21
percentage of BOLD signal
  Nicotine or satiety | 7.3 (15) | 6.3 (12)
  Placebo or abstinence | 6.2 (12) | .02 (8)

ADVERSE EVENTS:
Arm/Group | Nicotine, Placebo | Nicotine Withdrawal or Satiety
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/24
Other Adverse Events (participants affected / at risk) | 0/30 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No